CLINICAL TRIAL: NCT00444470
Title: Efficacy of Tranexamic Acid in Reducing Blood Loss in Adult Patients Having Major Spine Surgery
Brief Title: Safety of Tranexamic Acid in Reducing Bleeding in Adults Undergoing Spinal Surgery
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Jean Wong, MD, FRCPC, Department of Anesthesia, Toronto Western Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P.S.I. Grant No. 02-69
Record Dates: First submitted 2007-03-05; First posted 2007-03-07 (Estimated); Last update posted 2007-11-30 (Estimated); Status verified 2007-11

CONDITIONS: Spine Surgery
Keywords: tranexamic acid; safety; efficacy; spine surgery; spinal fusion and decompression; adult; perioperative; blood loss; bleeding; blood transfusion
MeSH Terms: conditions — Hemorrhage | interventions — Tranexamic Acid

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- A (Active Comparator): Active drug being tested in this study is Tranexamic Acid
  Interventions: Drug: Tranexamic acid
- B (Placebo Comparator): Normal saline was used as the Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Tranexamic acid — Eligible patients who have consented to be in the study and have been randomised to be in Arm "A" will receive 10 mg/kg of tranexamic acid, and then a continuous infusion of 1 mg/kg/hr of tranexamic acid.
  Other Names: Tranexamic acid is known by the brand name Cyclokapron
  Arms: A
Drug: Placebo — Eligible patients who have consented to be in the study and have been randomised to be in Arm "B" will receive 10 mg/kg of placebo followed by a continuous infusion of 1 mg/kg/hr of placebo.
  Other Names: Normal Saline is used as placebo
  Arms: B

SUMMARY:
Spinal fusion surgery can be associated with significant blood loss requiring allogeneic blood transfusion. Tranexamic acid is a synthetic amino acid with antifibrinolytic action that has been shown to reduce perioperative blood loss in patients undergoing cardiopulmonary bypass for cardiac bypass surgery, knee replacement and liver transplantation surgeries. The efficacy of antifibrinolytics for reduction of blood loss in major spine surgery has not been well studied in adult patients. The objective of this study is to determine the efficacy of tranexamic acid in reducing perioperative blood loss and blood transfusion in adults undergoing elective spinal fusion in a larger, multi-centered, randomized, double-blinded, placebo controlled trial.

DETAILED DESCRIPTION:
Spinal fusion can be associated with significant blood loss requiring allogeneic blood transfusion (ABT). Ongoing concerns about the costs, risks, and availability of allogeneic blood have prompted the implementation of multiple techniques (preoperative erythropoetin, autologous pre-donation, intra-operative blood salvage, and induced hypotension) to reduce the necessity of ABT. However, 28% of patients undergoing spinal fusion at the Toronto Western Hospital still receive ABT. Also, none of these modalities (with the exception of induced hypotension) actually reduce the amount of blood shed from the surgical wound; thus the severity of anemia is largely unaffected. Consequently, many of these patients can suffer from adverse effects of anemia postoperatively as well as potential complications from blood transfusions.

The underlying assumption of the proposed study is that excessive fibrinolysis occurs during spinal fusion surgery. This can result in increased and recurrent blood loss, which can exacerbate the significant amount of bleeding already associated with major spine surgery.

Tranexamic acid - an antifibrinolytic drug blocks the dissolution of hemostatic fibrin, which stabilizes fibrin structures, and thus may decrease blood loss secondary to increased fibrinolysis.

This research proposal will test the following hypotheses:

1. Tranexamic acid reduces the estimated perioperative blood loss in adult patients undergoing elective spinal fusion.
2. Tranexamic acid reduces the need for blood transfusion in adult patients undergoing elective spinal fusion.

This multi-centered trial will be valuable for establishing the efficacy and safety of tranexamic acid for reducing blood loss and allogeneic blood transfusion in adults having elective spinal fusion. Tranexamic acid is easy to administer, is relatively inexpensive, and has not been associated with significant adverse effects. If it is shown to be efficacious, it can be incorporated into routine clinical practice as part of the multi-modal perioperative blood conservation techniques currently used to reduce perioperative blood loss, transfusion and the risk of allogeneic blood transfusion.

ELIGIBILITY:
Inclusion Criteria:

* All adult patients (greater than 18 years old) undergoing elective posterior thoracic/lumbar instrumented spinal fusion.

Exclusion Criteria:

* Participation in another clinical trial
* Allergy to TA
* Spinal tumor/Intradural pathology
* Ankylosing spondylitis
* Acquired disturbances of color vision
* Preoperative anemia (Hb <110 in females, Hb <120 in males)
* Refusal of blood products (Jehovah's witnesses)
* Preoperative use of anticoagulant therapy - coumadin, heparin within 5 days of surgery
* Fibrinolytic disorders requiring intraoperative antifibrinolytic treatment
* Hematological disease (thromboembolic events, hemoglobinopathy, coagulopathy or hemolytic disease)
* Preoperative platelet count <150,000/cubic mm, INR>1.4, prolonged PTT
* Significant co-morbidities: Previous MI ; severe ischemic heart disease (NYHA Class III, IV) ; severe pulmonary disease ; chronic renal failure ; hepatic failure ; uncontrolled hypertension
* Pregnancy or lactation

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2003-02; Study Completion 2007-05 (Actual)

PRIMARY OUTCOMES:
Total perioperative blood loss | Measured intraoperatively and 24 hours postoperatively

SECONDARY OUTCOMES:
Incidence of autologous or allogeneic blood transfusion, including red blood cells and coagulation components, i.e., FFP and platelets | Administered during entire hospitalization
Other secondary outcomes will include hemoglobin concentration, fatigue and functional recovery, and duration of hospital stay. | Hemoglobin concentration will be measured pre-operatively, intraoperatively and on post-operative days 1-3. Fatigue questionnaire will be completed at the pre-operative admission, post-operative days 3 and 7, and after discharge at 6 weeks.

CONTACTS AND LOCATIONS:
Overall Officials: Jean Wong, MD, FRCPC, Principal Investigator — University Health Network, Toronto; Henry Ahn, MD, FRCPC, Study Director — Unity Health Toronto; Robert McBroom, MD, FRCPC, Study Director — Trillium Health Centre
Locations (3):
- Canada (3):
  - Trillium Health Centre, Mississauga, Ontario
  - St. Michael's Hospital, Toronto, Ontario
  - Department of Anesthesia and Orthopedics; Toronto Western Hospital, Toronto, Ontario